CLINICAL TRIAL: NCT07240519
Title: Vulvar Lichen Sclerosus: Expression of Inflammatory Markers in a Randomized Clinical Trial With Clobetasol Versus Laser
Brief Title: To Compare Inflammatory Biomarkers Before and After Treatment With Clobetasol or Fractional CO2 Laser, in Women With Histologically Confirmed Vulvar Lichen Sclerosus, Without Prior Corticosteroid Treatment.
Acronym: LASER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Andréa Cytryn, Principal investigator, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 52132021000005275
Record Dates: First submitted 2025-11-16; First posted 2025-11-21 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Vulvar Lichen Sclerosus
Keywords: CO2 laser; vulvar lichen sclerosus
MeSH Terms: conditions — Vulvar Lichen Sclerosus

STUDY DESIGN:
Intervention Model Description: Forty women will be randomized after histological confirmation of vulvar lichen sclerosus for one of the two arms. 20 women will be allocated to clobetasol group and 20 women will be allocated to CO2 laser group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Paricipants randomized for Clobetasol ointment group (Active Comparator): Participants in this group will apply clobetasol propionate 0.05% ointment to the vulvar affected area in an amount sufficient to cover the finger tip according to standard treatment protocol:
  every day in the first month every other day in the second month twice a week (for example: Mondays and Thursdays) in the third month
  Interventions: Device: Fractional microablative CO2 Laser
- Participants randomized for Fractional Carbon dioxide (CO2 ) laser group treatment (Experimental): Fractional microablative CO2 laser An anesthetic ointment provided by the principal investigator, applied on vulva skin, perineal area and vulvar vestibule 30 - 45 minutes before the Session of CO2 laser.
  Three sessions spaced four weeks apart, with instructions after each session, such as avoiding sexual intercourse for five days and using a product like petroleum jelly for relief for a few days.
  Interventions: Device: Fractional microablative CO2 Laser

INTERVENTIONS:
Device: Fractional microablative CO2 Laser — In this study the investigators use the laser device without any topic esteroid previous or during the period of laser sessions

SUMMARY:
The present study is a Clinical trial that compares clobetasol ointment versus Fractional CO2 laser for vulvar lichen sclerosus (VLE) treatment confirmed by histology, with no previous treatment. Lichen sclerosus is a chronic inflamatory disease that affects the vulvar skin in the majority of cases, generally in peri and post menopause. The main symptom is pruritus, along with dispareunia and vulvar pain. If not treated, it can leads to vulvar anatomy distortion and altough small, there is risk of neoplastic transformation towards pre cancer and invasive vulvar cancer. Clobetasol ointment is the standard treatment, but prolonged use can cause some adverse effects, such as thinning the skin, fungal infections, and exacerbation of symptoms. Forty participants are being randomized to clobetasol group, three months with reducing frequency and the other group of participants, to fractional dioxid carbon (CO2) laser for three sessions four weeks apart. At the beggining and three months after the completion of each treatment, a punch biopsy will be taken for every participant. The principal aim is to compare some inflamatory biomarkers before and after each treatment and compare them by imunohistoquemestry at Imunology and Imunogenetic Laboratory in Fiocruz, Rio de janeiro, Brazil.

Secondary outcomes include clinical response and changes in vulvar anatomy, assessed using the Sheinis & Selk questionnaire before and after each treatment, as well as the evaluation of some clinical aspects, such as improvement in itching, dyspareunia and appearance of the vulva, along with satisfaction with the treatment, using the Visual Analogue Scale (VAS) from 1 to 10.

With this study, the investigators want to know if fractional CO2 laser can reduce the inflammatory process and symptoms in vulvar lichen sclerosus such as itching, and if this could be an alternative treatment for this condition.

ELIGIBILITY:
Inclusion Criteria: Women older than 21 years; histological diagnostic of vulvar lichen sclerosus and no previous treatment with topic corticoesteroid

Exclusion Criteria: Women that don't agree in taking part of the study; other concomitant vulvar diseases; pre malignant vulvar disease HPV dependent and independent; previous pelvic radiotherapy

-

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-06-22 (Actual); Primary Completion 2025-09-10 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Evaluation and comparison of inflammatory biomarkers before and after treatment with clobetasol or CO2 laser. | Each participant will be monitored from registration, throughout treatment, and up to three months after the end of treatment.
  Before and after each of the two treatments, a vulvar punch biopsy will be performed. The fragment will then be analyzed using immunohistochemistry to assess changes in inflammatory biomarkers.
To evaluate the performance of CO2 laser in vulvar lichen sclerosus in relation to inflammatory skin markers and compare to clobetasol | From enrollment to a second biopsy 3 months after treatment
  In vulvar skin fragment obtained by punch biopsy, some inflammatory biomarkers such as TGF-β, INF-γ, VEGF, and IL-10 will be evaluated before and three months after the last laser session.
  The biomarkers will be quantified by immunohistochemistry at the Immunology and Immunogenetics Laboratory of Fiocruz.
  For the count, a compound optical microscope will be used, consisting of a 40x objective lens and a 10x grating eyepiece. The total number of cells positive for the marker being analyzed will be recorded in each field.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Cytryn, Master of Science in Health, Principal Investigator — Department of Gynecology, Institute of Gynecology, Federal University of Rio de janeiro
Locations (1):
- Institute of Gynecology of the Federal University of Rio de Janeiro, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Sociodemographic data such as age, race, marital status, education. Clnical data such as parity, mode of delivery, active or inactive sexual life, period of reproductive life and current contraception, presence of autoimmune diseases, comorbidities such as hypertension, diabetes, regular medications and smoking
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data becomes available 6 months after publication.

REFERENCES:
- [Result] Krause E, Neumann S, Maier M, Imboden S, Knabben L, Mueller MD, Kuhn A. LASER treatment in gynaecology -A randomized controlled trial in women with symptomatic lichen sclerosus. Eur J Obstet Gynecol Reprod Biol. 2023 Aug;287:171-175. doi: 10.1016/j.ejogrb.2023.06.003. Epub 2023 Jun 8. PMID 37352640
- [Result] Preti M, Vieira-Baptista P, Digesu GA, Bretschneider CE, Damaser M, Demirkesen O, Heller DS, Mangir N, Marchitelli C, Mourad S, Moyal-Barracco M, Peremateu S, Tailor V, Tarcan T, De EJB, Stockdale CK. The clinical role of LASER for vulvar and vaginal treatments in gynecology and female urology: An ICS/ISSVD best practice consensus document. Neurourol Urodyn. 2019 Mar;38(3):1009-1023. doi: 10.1002/nau.23931. Epub 2019 Feb 11. PMID 30742321
- [Result] Tasker F, Kirby L, Grindlay DJC, Lewis F, Simpson RC. Laser therapy for genital lichen sclerosus: A systematic review of the current evidence base. Skin Health Dis. 2021 Jun 15;1(3):e52. doi: 10.1002/ski2.52. eCollection 2021 Sep. PMID 35663131
- [Result] Burkett LS, Siddique M, Zeymo A, Brunn EA, Gutman RE, Park AJ, Iglesia CB. Clobetasol Compared With Fractionated Carbon Dioxide Laser for Lichen Sclerosus: A Randomized Controlled Trial. Obstet Gynecol. 2021 Jun 1;137(6):968-978. doi: 10.1097/AOG.0000000000004332. PMID 33957642
- [Result] Filippini M, Sozzi J, Farinelli M, Verdelli A. Effects of Fractional CO2 Laser Treatment on Patients Affected by Vulvar Lichen Sclerosus: A Prospective Study. Photobiomodul Photomed Laser Surg. 2021 Dec;39(12):782-788. doi: 10.1089/photob.2021.0053. PMID 34878932
- [Result] Singh N, Ghatage P. Etiology, Clinical Features, and Diagnosis of Vulvar Lichen Sclerosus: A Scoping Review. Obstet Gynecol Int. 2020 Apr 21;2020:7480754. doi: 10.1155/2020/7480754. eCollection 2020. PMID 32373174
- [Result] Farrell AM, Dean D, Millard PR, Charnock FM, Wojnarowska F. Cytokine alterations in lichen sclerosus: an immunohistochemical study. Br J Dermatol. 2006 Nov;155(5):931-40. doi: 10.1111/j.1365-2133.2006.07414.x. PMID 17034521
- [Result] Krapf JM, Mitchell L, Holton MA, Goldstein AT. Vulvar Lichen Sclerosus: Current Perspectives. Int J Womens Health. 2020 Jan 15;12:11-20. doi: 10.2147/IJWH.S191200. eCollection 2020. PMID 32021489
- See also: Related Info — https://www.issvd.org